CLINICAL TRIAL: NCT02486237
Title: Complications in Central American Diabetic Patients: Historic Cohort
Status: Completed | Type: Observational
Sponsor: Clínica Los Yoses (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Chih Hao Chen Ku, MD, Clínica Los Yoses
Other Study IDs: 001
Record Dates: First submitted 2015-06-22; First posted 2015-07-01 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes mellitus; complications; prevalence
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 2 diabetes mellitus: Type 2 diabetes mellitus patients, no intervention is performed besides usual clinical practice
  Interventions: Other: None, observational study

INTERVENTIONS:
Other: None, observational study — None, it is an observational study

SUMMARY:
Retrospective, observational study to determine the prevalence of complications in Central American diabetic patients.

DETAILED DESCRIPTION:
This is retrospective observational study aimed to determine the prevalence of complications in Central American diabetic patients. Patients included are treated in the usual outpatient practice setting and we will try to determine the prevalence of diabetic complications in these patients.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus diagnosed between 2004 and 2009
* seen by the attending physician for the first time between January and December 2009.
* male or female patients between 18 and 80 years

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with type 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with microvascular and cardiovascular complications | up to 10 years

SECONDARY OUTCOMES:
Number of participants with at least one episode of hypoglycemia | up to 10 years
Number of patients with microvascular and cardiovascular complications stratified by their glucose control | up to 10 years
Number of patients with microvascular and cardiovascular complications stratified by blood pressure control | up to 10 years
Number of patients with microvascular and cardiovascular complications stratified by cholesterol levels | up to 10 years
Number of patients with microvascular and cardiovascular complications stratified by diabetes pharmacologic treatment | up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Chih Hao Chen Ku, MD, Principal Investigator — Clínica Los Yoses
Locations (8):
- Costa Rica (2):
  - Hospital CIMA, San José, Provincia de San José
  - Clínica Los Yoses, San Pedro, Provincia de San José
- El Salvador (3):
  - Centro Panamericano de Ojos, San Salvador, San Salvador Department
  - INSACOR, San Salvador, San Salvador Department
  - Medicentro La Esperanza, San Salvador, San Salvador Department
- Guatemala (2):
  - Clínica 1005, Guatemala City, Departamento de Guatemala
  - Prevención en Salud S.A, Guatemala City, Departamento de Guatemala
- Honduras Medical Center, Tegucigalpa, Francisco Morazán Department, Honduras

IPD SHARING:
Plan to Share IPD: Undecided